CLINICAL TRIAL: NCT02073903
Title: The Use of Dual-handset Interpreter Phones in an Inpatient Setting to Improve Communication With Limited English Proficiency Patients at MSKCC
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-042
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Inpatients With Limited English Proficiency
Keywords: dual handset interpreter phones; communication; 14-042
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LEP inpatients and their providers: This is a feasibility project with the goal of improving communication between limited English proficiency (LEP )inpatients and their providers. Quantitative data will be obtained via two surveys: a patient survey to assess patients' feedback on the effectiveness of the communication during their hospital stay and their understanding of their medical care, and a provider survey to assess the handset's impact on the effectiveness of the communication. From this data we will be able to assess patient and provider communication effectiveness with both the current various practices at MSKCC and the new intervention.
  Interventions: Behavioral: Patient Survey; Behavioral: Provider Survey

INTERVENTIONS:
Behavioral: Patient Survey
Behavioral: Provider Survey

SUMMARY:
The purpose of this study is to introduce new technology and interpreter practices in the inpatient setting at MSKCC. We plan to install dual handset phones at the bedsides of limited English proficiency (LEP) patients and to assess the impact on both patient and physician communication effectiveness with this technology.

DETAILED DESCRIPTION:
During the first 5-6 weeks of the study standard of care will be conducted as usual practice by the medicine teams at MSKCC. It is expected that during that time they will care for at least 20 LEP patients who meet our inclusion criteria. There are no specific target numbers for any of the included languages. During the following 5-6 weeks, the phones will be installed by the 10 house-staff teams and approximately an additional 20 LEP patients who meet the protocol inclusion criteria will be enrolled. Therefore, in the first half of this study about 20 LEP patients and 40 practitioners (two practitioners per LEP patient) will provide data and the same numbers will account for the second half of the study after the intervention is instituted. There will be no randomization of patients or physicians. The only data that will be analyzed are those questions from the surveys to assess communication effectiveness with LEP patients. The number of patients who are interviewed will depend on MSKCC inpatient census at the time of study.

ELIGIBILITY:
Inclusion Criteria:

* LEP patients identified by the Department of Interpreter Services at MSKCC admitted to the Hepatobiliary surgery service, the Colorectal Surgery service the GMT surgery service, GI, GU, Breast, General Medicine, Leukemia, or Lymphoma services with a primary language of Spanish, Russian, or Chinese.
* LEP patients who are expected to have at least a two days hospital course.
* Patients who are alert and oriented to person, place, and time as determined by the medical doctor taking care of the patient
* Patients who are willing to participate and complete the survey
* Patients whose physicians and nurses are willing to participate
* Only persons ≥ 18 will be included and there will be no children.
* Providers must be willing to participate and complete the survey
* TY interns cannot complete provider surveys

Exclusion Criteria:

* Patients on contact isolation
* Patients who previously completed the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient Support Services will generate a daily list of inpatients that prefer to communicate in a language other than English.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Patient communication effectiveness | 1 year
  with the dual handset phones assessed by the survey

SECONDARY OUTCOMES:
Physician and nurse communication effectiveness | 1 year
  with the dual handset phones assessed by the survey

CONTACTS AND LOCATIONS:
Overall Officials: Chhavi Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/